CLINICAL TRIAL: NCT01009658
Title: Effect of Monosodium Glutamate on Upper Gastrointestinal Tract Motility
Brief Title: MSG and Gastrointestinal Motility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gunma University (Other)
Responsible Party: Principal Investigator, Hiroko Hosaka, MD, Gunma University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: GU-696; GU-CT 696
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Gastroesophageal Reflux
Keywords: Gastrointestinal motility; Gastroesophageal reflux; Gastric emptying; Sodium glutamate; Lower esophageal sphincter
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Sodium Glutamate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- MSG first (Active Comparator)
  Interventions: Dietary Supplement: Monosodium glutamate
- NaCl first (Placebo Comparator)
  Interventions: Dietary Supplement: Sodium chloride

INTERVENTIONS:
Dietary Supplement: Monosodium glutamate — Oral intake of 2.0 g of monosodium glutamate on the examination day and 0.6 g of sodium chloride on the other examination day.
  Arms: MSG first
Dietary Supplement: Sodium chloride — Oral intake of 0.6 g of sodium chloride on the examination day and 2.0 g of monosodium glutamate on the other examination day.
  Arms: NaCl first

SUMMARY:
The purpose of this study is to clarify the physiological function of sodium glutamate by measuring its effect on upper GI motility ( gastric emptying).

DETAILED DESCRIPTION:
Amino acids such as monosodium glutamate are known to stimulate both endocrine and exocrine secretion. In addition, there is a report that oral intake of glutamate evokes the activation of vagal afferent nerves in the rat. Thus, such amino acids are thought to be influential in the process of digestion and absorption.

. To investigate the effect of monosodium glutamate on gastrointestinal motility, we planned a single-blind randomized study. The participants will take either monosodium glutamate or sodium chloride before the first examination of upper GI motility and the other agent before the second examination. The order of intake will be randomized by the envelope method.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Must not have digestive symptoms
* Must not eat within six hours of study participation

Exclusion Criteria:

* Regular medications for the gastrointestinal tract
* Previous Helicobacter pylori infection
* Previous abdominal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-12; Primary Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Gastric emptying | 0-5 hours
  half emptying time

CONTACTS AND LOCATIONS:
Locations (1):
- Gunma university hospital, Maebashi, Gunma, Japan